CLINICAL TRIAL: NCT03107286
Title: Biokinetics Study for Tc-99m MAG3 Dose Reduction in Pediatric Molecular Imaging
Brief Title: Biokinetics Study for Tc-99m MAG3 in Pediatric Molecular Imaging
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Johns Hopkins University (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Frederic Fahey, Professor of Radiology, Boston Children's Hospital
Other Study IDs: IRB-P00025086_3
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Tc-99m MAG3: Children ages 1-6 years old will be eligible to participate. Routine imaging is performed immediately as a dynamic acquisition with 80 frames over 20 min. (15 s per frame). Subjects in each age group will be additionally imaged 2-3 h post-administration. It is important to note that the patient volunteers will not receive any additional radiation exposure for inclusion in this study. They are only being ask to allow imaging at one additional time point.
  Interventions: Drug: Tc-99M-MAG3; Other: Modification in acquisition protocol

INTERVENTIONS:
Drug: Tc-99M-MAG3 — Participants will be asked to be imaged at an additional time point during a nuclear medicine study using Tc-99m MAG3
Other: Modification in acquisition protocol — Participants will be asked to be imaged at an additional time point.

SUMMARY:
The radiation exposure resulting from medical imaging is a topic of some concern. Nuclear medicine provides potentially life-saving information regarding physiological processes, and is of particular value in children where the rapid and unequivocal diagnosis of pathological concerns is essential for the health of these patients. The overall objective of this investigation is to optimize pediatric patient absorbed dose by keeping it as low as possible while maintaining excellent diagnostic quality of nuclear medicine images. This is particularly important since children are at increased risk due to the enhanced radiosensitivity of their tissues and the longer time-period over which radiation effects may manifest. Current dosimetric estimations in children are based on either animal biokinetic or pharmacokinetic data from adults due to paucity of data that exists for children. This situation will be improved through the following specific aims:

* Collect image-based pharmacokinetic (PK) data from patient volunteers in different age groups scheduled for routine nuclear medicine studies for Tc-99m mercaptoacetyltriglycine (MAG3), a radiopharmaceutical commonly used in pediatric nuclear medicine
* Pool and analyze the data for different age groups for each radiopharmaceuticals and
* Generate biokinetic models to be used in subsequent dosimetric models for the optimization of pediatric nuclear medicine procedures.

Since inadequate pharmacokinetic data currently exist in these patients, the investigators will use the data acquired in this study to establish PK models applicable to different age categories. Data on the pharmacokinetics of agents used in pediatric nuclear medicine are almost completely lacking. Internationally adopted dose coefficients (mSv/MBq) for pediatric nuclear medicine make age-dependent adjustments only for patient size and anatomical differences, while time-dependent kinetics from adult PK models are assumed due to the lack of kinetic data for children. The data obtained from this study will make it possible for the first time to determine how the PK in pediatric patients differs from adults. This will be done for Tc-99m MAG3, a radiopharmaceutical commonly used for pediatric nuclear medicine imaging. The overall hope is that results will allow the molecular imaging community to implement pediatric dose-reduction approaches that substantially improve upon current guidelines pointing to future technological advances that could yield even greater dose-reduction while simultaneously improving diagnostic image quality.

DETAILED DESCRIPTION:
The overall objective of this investigation is to optimize pediatric patient absorbed dose by keeping it as low as possible while maintaining and even improving the diagnostic quality of nuclear medicine images. Current dosimetric estimations in children are based on either animal biokinetic or pharmacokinetic data from adults. This is due to paucity of data that exists specifically for children. This situation will be improved through the following specific aims:

* Collect imaging-based pharmacokinetic (PK) data from patient volunteers in different age groups scheduled for selected, routine nuclear medicine studies for Tc-99m MAG3, a radiopharmaceutical commonly used in pediatric nuclear medicine
* Pool and analyze the data for different age groups for each radiopharmaceuticals and
* Generate biokinetic models to be used in subsequent dosimetric models for the optimization of pediatric nuclear medicine procedures.

Pediatric absorbed dose estimates that are typically reported apply adult PK data with pediatric variations in body size and anatomy but not for differences in physiology between children and adults. Depending on the diagnostic agent, such differences can be of greater impact than anatomical differences. The investigators will acquire image data that will allow us to develop PK models for Tc-99m mercaptoacetyltriglycine (MAG3), a radiopharmaceutical routinely used in pediatric nuclear medicine for renal imaging. Patients undergoing standard of care imaging will be asked to consent to being imaged at one additional time point, either prior or subsequent to the time typical for clinical imaging. No patient will be asked to undergo more than one additional imaging time-point.

It is important to note that the patient volunteers will not receive any additional radiation exposure for inclusion in this study. They are only being ask to allow imaging at an additional time point.

Children ages 1-6 years old will be eligible to participate. Routine imaging is performed immediately as a dynamic acquisition with 80 frames over 20 min. (15 s per frame). Subjects in each age group will be additionally imaged 2-3 h post-administration.

The additional imaging will occur on the day of the clinically indicated procedure. Other than that, there is no timeline associated with this study.

Image data acquired from the subjects will be analyzed by the principle investigator and by colleagues at Johns Hopkins University and the University of Florida. Regions of interest will be defined around pertinent target organs and tissues and the count data recorded. The specific target organs will depend on the particular radiopharmaceutical. The data for each age range and time point will be pooled, normalized and fit to models describing the pharmacokinetics. The resultant models will be evaluated for age-based variations in the PK data and compared to existing, published models based on adult data to evaluated age based differences. Lastly, the impact that the more accurate PK has on dosimetric estimates of patients of different ages will be analyzed.

The number of subjects required at each time point will be determined using nonlinear mixed effects modeling software to model the data and adjust for covariates. The likelihood ratio test based on the objective function value (OFV) will be used to estimate PK parameters for varying doses and ages using a Bayesian approach. The proposed sample size plan with subjects imaged at different time points is predicated on the Monte Carlo Mapped Power (MCMP) method to achieve 80% power for detecting age and dose effects and robust coverage in estimating individual PK parameters. It is expected that there will be 5-10 subjects per age group depending on the statistical requirements as described above.

ELIGIBILITY:
Inclusion Criteria:

* All patients within the specified age ranges scheduled at Boston Children's Hospital for a nuclear medicine study utilizing Tc-99m MAG3 will be eligible to volunteer for inclusion in this study. It is also essential that inclusion does not compromise the potential of acquiring the clinically indicated image acquisition.

Exclusion Criteria:

* Inability to be imaged at the additional time point without the need for sedation or anesthesia

Ages: 9 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients within the specified age ranges scheduled at Boston Children's Hospital for a nuclear medicine study utilizing Tc-99m MAG3 will be eligible to volunteer for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Radioactivity in target organs at various time points | 6 hours
  The target-organ radioactivity measurements will be used to estimate the time-integrated activity in the target organs, hopefully leading to better estimates of absorbed dose to patients of different ages.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic H Fahey, DSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data, with all protected patient information removed, will be shared with collaborators at Johns Hopkins University and the University of Florida. In particular, anonymized nuclear medicine image data will be shared for analysis.

REFERENCES:
- [Background] Fahey FH, Goodkind AB, Plyku D, Khamwan K, O'Reilly SE, Cao X, Frey EC, Li Y, Bolch WE, Sgouros G, Treves ST. Dose Estimation in Pediatric Nuclear Medicine. Semin Nucl Med. 2017 Mar;47(2):118-125. doi: 10.1053/j.semnuclmed.2016.10.006. Epub 2016 Nov 9. PMID 28237000
- [Background] Treves ST, Gelfand MJ, Fahey FH, Parisi MT. 2016 Update of the North American Consensus Guidelines for Pediatric Administered Radiopharmaceutical Activities. J Nucl Med. 2016 Dec;57(12):15N-18N. No abstract available. PMID 27909182
- [Background] Fahey FH, Ziniel SI, Manion D, Baker A, Treves ST. Administered Activities in Pediatric Nuclear Medicine and the Impact of the 2010 North American Consensus Guidelines on General Hospitals in the United States. J Nucl Med. 2016 Sep;57(9):1478-85. doi: 10.2967/jnumed.116.172148. Epub 2016 Apr 7. PMID 27056617
- [Background] Grant FD, Gelfand MJ, Drubach LA, Treves ST, Fahey FH. Radiation doses for pediatric nuclear medicine studies: comparing the North American consensus guidelines and the pediatric dosage card of the European Association of Nuclear Medicine. Pediatr Radiol. 2015 Apr;45(5):706-13. doi: 10.1007/s00247-014-3211-x. Epub 2014 Nov 1. PMID 25367355